CLINICAL TRIAL: NCT03133169
Title: Erythrocyte Glutamine Level Relation to Pulmonary Hypertension Risk in Beta Thalassemia Major Children in Assiut University Children Hospital
Brief Title: Erythrocyte Glutamine Level Relation to Pulmonary Hypertension Risk in Beta Thalassemia Major Children
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Sami, Pediatric Resident, Assiut University
Other Study IDs: GlnThalassemia
Record Dates: First submitted 2017-04-15; First posted 2017-04-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Thalassemia in Children; Pulmonary Hypertension; Hemolysis
Keywords: Thalassemia; Glutamine/glutamate ratio; Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Hemolysis; Thalassemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- on chelation: patients with B-thalassemia major samples of which will be examined for renal and liver function, Erythrocyte Glutamine level, ferritin level and complete blood picture. Also Echo will be done for measuring the Tricuspid regurge velocity.
  group 1: cases on chelation: deferasirox 500mg oral tablet with initial dose 20 mg/kg guided by ferritin level
  Diagnostic Test: blood sample
  Diagnostic Test: Tricuspid regurge velocity
  Interventions: Diagnostic Test: blood sample; Diagnostic Test: Tricuspid regurge velocity
- No chelation: group 2: cases without chelation
  Diagnostic Test: blood sample
  Diagnostic Test: Tricuspid regurge velocity
  Interventions: Diagnostic Test: blood sample; Diagnostic Test: Tricuspid regurge velocity
- splenectomy: group 3: cases with splenectomy
  Diagnostic Test: blood sample
  Diagnostic Test: Tricuspid regurge velocity
  Interventions: Diagnostic Test: blood sample; Diagnostic Test: Tricuspid regurge velocity
- no splenectomy: group 4: cases without splenectomy Diagnostic Test: blood sample Diagnostic Test: Tricuspid regurge velocity
  Interventions: Diagnostic Test: blood sample; Diagnostic Test: Tricuspid regurge velocity

INTERVENTIONS:
Diagnostic Test: blood sample — blood sample for measuring liver and kidney function, CBC, ferritin level and erythrocyte glutamine level
Diagnostic Test: Tricuspid regurge velocity — Tricuspid regurge velocity will be measured by doppler echocardiography denoting the pulmonary hypertension risk in children

SUMMARY:
The study will investigate the relation between erythrocyte glutamine/glutamate ratio and pulmonary hypertension risk in Egyptian thalassemic children in Assiut University Children Hospital

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Thalassemia.
* PH risk documented by doppler echocardiography, defined as tricuspid regurge velocity (TRV) equal to or greater than 2.5 m/s

Exclusion Criteria:

* Acute crisis or hospitalization within 1 month of enrollment
* Hepatic dysfunction (SGPT greater than 3X normal)
* Renal dysfunction (Creatinine greater than 2X normal)
* Patients on sildenafil (Viagra), calcium channel blockers or other drugs for the control of PH.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Upper Egypt thalassemic children aged 10-18 years old attending Assiut University Children Hospital.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Erythrocyte glutamine level | 2 months
  marker for oxidative stress
Tricuspid regurge velocity | 2 months
  Measures the risk of pulmonary hypertension

SECONDARY OUTCOMES:
Plasma glutamine level | 2 months
  Assess the glutamine level at each visit
Liver function tests | 2 months
  Evaluates the state of liver
Renal function tests | 2 months
  Evaluates the state of kidney
Ferritin level | 2 months
  measuring the iron overload

CONTACTS AND LOCATIONS:
Overall Officials: Fahim M Fahim, PhD, Principal Investigator — Children Hospital, Assiut University; Fatma S AbdElshafi, bachelor's, Principal Investigator — Children Hospital, Assiut University; Eman F. Mohamed, PhD, Principal Investigator — Children Hospital, Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] Morris CR, Kuypers FA, Kato GJ, Lavrisha L, Larkin S, Singer T, Vichinsky EP. Hemolysis-associated pulmonary hypertension in thalassemia. Ann N Y Acad Sci. 2005;1054:481-5. doi: 10.1196/annals.1345.058. PMID 16339702
- [Background] Morris CR, Vichinsky EP. Pulmonary hypertension in thalassemia. Ann N Y Acad Sci. 2010 Aug;1202:205-13. doi: 10.1111/j.1749-6632.2010.05580.x. PMID 20712794
- [Background] Walter PB, Fung EB, Killilea DW, Jiang Q, Hudes M, Madden J, Porter J, Evans P, Vichinsky E, Harmatz P. Oxidative stress and inflammation in iron-overloaded patients with beta-thalassaemia or sickle cell disease. Br J Haematol. 2006 Oct;135(2):254-63. doi: 10.1111/j.1365-2141.2006.06277.x. PMID 17010049
- [Background] Morris CR. Mechanisms of vasculopathy in sickle cell disease and thalassemia. Hematology Am Soc Hematol Educ Program. 2008:177-85. doi: 10.1182/asheducation-2008.1.177. PMID 19074078
- [Background] Kuypers FA. Membrane lipid alterations in hemoglobinopathies. Hematology Am Soc Hematol Educ Program. 2007:68-73. doi: 10.1182/asheducation-2007.1.68. PMID 18024611
- [Background] Fung EB, Harmatz P, Milet M, Ballas SK, De Castro L, Hagar W, Owen W, Olivieri N, Smith-Whitley K, Darbari D, Wang W, Vichinsky E; Multi-Center Study of Iron Overload Research Group. Morbidity and mortality in chronically transfused subjects with thalassemia and sickle cell disease: A report from the multi-center study of iron overload. Am J Hematol. 2007 Apr;82(4):255-65. doi: 10.1002/ajh.20809. PMID 17094096
- [Background] Machado RF, Gladwin MT. Pulmonary hypertension in hemolytic disorders: pulmonary vascular disease: the global perspective. Chest. 2010 Jun;137(6 Suppl):30S-38S. doi: 10.1378/chest.09-3057. PMID 20522578
- [Background] Janda S, Shahidi N, Gin K, Swiston J. Diagnostic accuracy of echocardiography for pulmonary hypertension: a systematic review and meta-analysis. Heart. 2011 Apr;97(8):612-22. doi: 10.1136/hrt.2010.212084. Epub 2011 Feb 25. PMID 21357375
- [Background] De Castro LM, Jonassaint JC, Graham FL, Ashley-Koch A, Telen MJ. Pulmonary hypertension associated with sickle cell disease: clinical and laboratory endpoints and disease outcomes. Am J Hematol. 2008 Jan;83(1):19-25. doi: 10.1002/ajh.21058. PMID 17724699
- [Background] Anthi A, Machado RF, Jison ML, Taveira-Dasilva AM, Rubin LJ, Hunter L, Hunter CJ, Coles W, Nichols J, Avila NA, Sachdev V, Chen CC, Gladwin MT. Hemodynamic and functional assessment of patients with sickle cell disease and pulmonary hypertension. Am J Respir Crit Care Med. 2007 Jun 15;175(12):1272-9. doi: 10.1164/rccm.200610-1498OC. Epub 2007 Mar 22. PMID 17379852
- [Background] Hebbel RP. Reconstructing sickle cell disease: a data-based analysis of the "hyperhemolysis paradigm" for pulmonary hypertension from the perspective of evidence-based medicine. Am J Hematol. 2011 Feb;86(2):123-54. doi: 10.1002/ajh.21952. PMID 21264896
- [Background] Morris CR. Vascular risk assessment in patients with sickle cell disease. Haematologica. 2011 Jan;96(1):1-5. doi: 10.3324/haematol.2010.035097. No abstract available. PMID 21193426
- [Background] Mok E, Hankard R. Glutamine supplementation in sick children: is it beneficial? J Nutr Metab. 2011;2011:617597. doi: 10.1155/2011/617597. Epub 2011 Nov 14. PMID 22175008
- [Background] Xu H, Pearl RG. Effect of l-glutamine on pulmonary hypertension in the perfused rabbit lung. Pharmacology. 1994 Apr;48(4):260-4. doi: 10.1159/000139188. PMID 8177911
- [Background] Morris CR, Suh JH, Hagar W, Larkin S, Bland DA, Steinberg MH, Vichinsky EP, Shigenaga M, Ames B, Kuypers FA, Klings ES. Erythrocyte glutamine depletion, altered redox environment, and pulmonary hypertension in sickle cell disease. Blood. 2008 Jan 1;111(1):402-10. doi: 10.1182/blood-2007-04-081703. Epub 2007 Sep 11. PMID 17848621
- [Background] Niihara Y, Matsui NM, Shen YM, Akiyama DA, Johnson CS, Sunga MA, Magpayo J, Embury SH, Kalra VK, Cho SH, Tanaka KR. L-glutamine therapy reduces endothelial adhesion of sickle red blood cells to human umbilical vein endothelial cells. BMC Blood Disord. 2005 Jul 25;5:4. doi: 10.1186/1471-2326-5-4. PMID 16042803
- [Background] Machado RF, Farber HW. Pulmonary hypertension associated with chronic hemolytic anemia and other blood disorders. Clin Chest Med. 2013 Dec;34(4):739-52. doi: 10.1016/j.ccm.2013.08.006. Epub 2013 Oct 17. PMID 24267302